CLINICAL TRIAL: NCT02678546
Title: Traditional Chinese Medicine Constitution Study and the Diagnosis and Treatment of Chronic Disease in Taiwan Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH104-REC3-097
Record Dates: First submitted 2016-01-12; First posted 2016-02-09 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Autoimmune Rheumatologic Disease; Kidney Disease; Endocrine, Metabolic or Nutritional Diseases or Conditions
Keywords: Traditional Chinese Medicine
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients in outpatients departments: patients from outpatients departments in teaching hospital
  Interventions: Other: Other
- General: participants from center of continuing education in China Medical University

INTERVENTIONS:
Other: Other — case review of diagnosed disease
  Groups: patients in outpatients departments

SUMMARY:
Several questionnaires have been developed for clinical research in Traditional Chinese Medicine. The objective of this study is to evaluate the consistency and relevance of two questionnaires, the Constitution in Chinese Medicine Questionnaire (CCMQ) and the Body Constitutions Questionnaire (BCQ).

DETAILED DESCRIPTION:
Aim: Several questionnaires have been developed for clinical research in Traditional Chinese Medicine. The objective of this study is to evaluate the consistency and relevance of two questionnaires, the Constitution in Chinese Medicine Questionnaire (CCMQ) and the Body Constitutions Questionnaire (BCQ).

Method: Between December 2015 and December 2016, a sample of 150 participants aged above 20 years from the Chinese Medical University "elder college" curriculum and outpatients at the Hospital in Taichung, Taiwan, will be interviewed to complete both questionnaires based on subjective symptoms in a 3-d interval. There are three common patterns of body constitutions in CCMQ and BCQ: gentleness/plain, Ying-deficiency, and Yang-deficiency. As for other body constitutions, Qi-deficiency, phlegm-dampness, dampness-heat, blood-stasis, Qi-depression, and special diathesis are described only in CCMQ, while stasis is a feature only defined in BCQ. Average and standard deviation will be used to describe the measurement scores of the questionnaires and the percentages of constitution distribution. Statistical analysis of the Kappa value, Pearson Chi-Square, odds ratio, and Pearson's correlation coefficient would be employed to examine the consistency and association between the two questionnaires.

Expected result: The investigators hope to 1) describe the constitution profile of the study population; 2) assess the consistency between two questionnaires; and 3) examine the associations between CCMQ and demographic life style factors.

ELIGIBILITY:
Inclusion Criteria:

* people above 20 years old

Exclusion Criteria:

* people who cannot understand the description of questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Population from Center of Continuing Education in China Medical University and patients from China Medical University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the measure patterns of the Constitution in Chinese Medicine Questionnaire (CCMQ) | 1 month
the measure patterns of the Body Constitutions Questionnaire (BCQ) | 1 month

SECONDARY OUTCOMES:
the association between measure patterns of CCMQ and demographic life style factors | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hen-Hong Chang, M.D.,Ph.D., Principal Investigator — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No